CLINICAL TRIAL: NCT04783129
Title: Multidisciplinary Health Educational Program Based on Centered People Care Model in Parkinson's Disease: Comparison Between Remote and Face-to-face Delivery
Brief Title: Multidisciplinary Health Educational Program Based on Centered People Care Model in Parkinson's Disease
Acronym: AMPARO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMPARO study
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Telehealth; People centered-care; Quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Stratified, single-blind, parallel-group, randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: All groups will be assessed before (baseline), and after the end of the intervention by a blinded examiner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face group (Experimental): Face-to-face group (FFG), in which participants, in groups of 10 persons, followed a multidisciplinary health education program composed of 10 monthly face-to-face lectures
  Interventions: Other: Education program based on 10 monthly lectures
- Remote group (Active Comparator): Remote group (RG), in which individuals followed 10 monthly remote lectures
  Interventions: Other: Education program based on 10 monthly lectures
- Control group (Sham Comparator): Control group (CG), in which participants followed no education program (lectures)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Education program based on 10 monthly lectures — The education program consist of 10 lectures on the management of motor and non-motor alterations associate with PD will be offered by a nurse, physiotherapist, occupational therapist, speech therapist, neurologist, lawyer, nutritionist, and psychologist.
  Arms: Face-to-face group; Remote group
Other: No intervention — Participants will follow no education program (lecture) and will be instructed to follow their usual routine for the treatment of the disease
  Arms: Control group

SUMMARY:
The objective of this study is to compare the effects of two similar long-term interprofessional programs, one of them delivers by in-person classes, and another delivers by online classes on the quality of life of people with Parkinson's.

Method: People with PD will be randomized into 3 groups: (1) Face-to-face group, in which participants, in groups of 10 persons, followed a multidisciplinary health education program composed of 10 monthly face-to-face lectures; (2) Remote group, in which individuals followed the same lectures delivered by online; and (3) Control group, in which participants followed no lecture. The participants will be evaluated before (BED) and after (ABP) the education program conclusion (10 lectures). Health quality of life was adopted as a primary outcome. Independence in daily living activities, motor and non-motor symptoms severity, and global cognitive capacity was adopted as secondary measures, Besides, all participants will be asked to answer a survey to evaluate the knowledge improvement of key learning points of lectures. The results will be analyzed by ANOVA for repeated measures.

DETAILED DESCRIPTION:
Parkinson's disease is a large cause of disability worldwide. The complex combination of motor and non-motor symptoms brings an increasing impairment in functionality and, consequently, a progressively decrease in the quality of life of the people living with PD and their families. The World Health Organization (WHO) recommends that for health care, especially in chronic diseases, care should be centered on the person (people-centered care). This model enlarges the focus on biological aspects, including psychological and social aspects, building a multidimensional perspective on an individual, which can only be reached by integrated and interprofessional care.

According to this model, education is crucial to empower the person to occupy an active role in the health process, gaining greater control over decisions and actions affecting their health. Patient empowerment has been associated with positive health and clinical outcomes, including improved disease management, effective use of health services, improved health status, and medication adherence. However, there are several barriers for participants to attending this kind of program. Reasons for nonparticipation include mobility-reducing physical health issues, time constraints, distance, insufficient funds, lack of respite care if caring for someone else, and transportation. Thus, using a home-based video class may be one opportunity to reduce these known barriers and improve the accessibility of education programs. This delivery strategy can be beneficial for no high-income countries.

Objective: The objective of this study is to compare the effects of two similar long-term interprofessional programs, one of them delivers by in-person classes, and another delivers by online classes on the quality of life of people with Parkinson's.

Method: People with a confirmed diagnosis of Idiopathic Parkinson's disease, in stage 1-4 of disease evolution according to Hoehn and Yahr classification will be randomized into 3 groups: (1) Face-to-face group (FFG), in which participants, in groups of 10 persons, followed a multidisciplinary health education program composed of 10 monthly face-to-face lectures; (2) Remote group (RG), in which individuals followed the same lectures delivered by online; and (3) Control group (CG), in which participants followed no lecture. People who have severe cognitive decline and uncorrected visual or hearing impairment will be excluded. Participants from both groups will be instructed to follow their usual routine for the treatment of the disease. The lectures on the management of motor and non-motor alterations associate with PD will be offered by a nurse, physiotherapist, occupational therapist, speech therapist, neurologist, lawyer, nutritionist, and psychologist. The participants will be evaluated before (BED) and after (ABP) the education program conclusion (10 lectures). Health quality of life, adopted as a primary outcome, will be evaluated by Parkinson´s disease questionnaire 39 (PDQ-39). The independence in daily living activities, motor and non-motor symptoms severity, and global cognitive capacity, adopted as secondary measures, will be evaluated by Unified Parkinson´s disease rating scale (UPDRS) and Montreal Cognitive Assessment (MoCA), respectively. Besides, all participants will be asked to answer a survey to evaluate the knowledge improvement of key learning points of lectures. The survey consisted of 20 questions (2 per lecture) where the minimum level (score 0) indicated the absence of knowledge and maximal level (score 5) indicated the full understanding of lectures' key points. The results will be analyzed by ANOVA for repeated measures considering as factor group (FFG, RG, CG) and assessment points (BED, AEP).

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Idiopathic Parkinson's disease Must have acess to internet.

Exclusion Criteria:

Severe cognitive decline Severe visual impairment Severe hearing impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in Health related Quality of life | baseline and immediately after the end of intervention
  Parkinson´s disease questionnaire 39 (PDQ-39), PDQ-39 is a widely used and acknowledged disease-specific, self-reported questionnaire. It contains 39 questions covering eight distinct domains: mobility, activities of daily living, emotional wellbeing, stigma, social support, cognition, communication, and bodily discomfort. The score for each question ranges from 0 to 4 points, with higher scores indicating higher levels of perceived problems. A change of ≥1.6 points on the PDQ-39 total score after 6 months represents a minimally clinically important difference

SECONDARY OUTCOMES:
Change in Unifed Parkinson's Disease Rating Scale scores | baseline and immediately after the end of intervention
  UPDRS - Part I: Non-Motor Experiences of Daily Living which has six rater-based items and seven for patient self-assessment; UPDRS - Part II: Motor experiences of daily living, with 13 patient-based items; UPDRS - Part III: Motor examination, 18 items based on clinical tests. Each item scores from 0 (normal) to 4 (severe) and total scores are obtained from the sum of the corresponding item scores for each part.
Change in Montreal Cognitive Assessment scores | baseline and immediately after the end of intervention
  Montreal Cognitive Assessment (MoCA): The 30-point designed to detect mild cognitive impairment and reportedly takes <10 min to administer with scores <26 defined as abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No